CLINICAL TRIAL: NCT05122364
Title: Telerehabilitation and Telecoaching of Parents of Cochlear Implanted Children at Sohag University Hospital
Brief Title: Telerehabilitation & Telecoaching of Parents of Cochlear Implanted Children at Sohag University Hospital
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, hadeel elsayed awad, Assistant lecturer, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 987321654
Record Dates: First submitted 2021-10-30; First posted 2021-11-16 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Cochlear Implantation; Hearing Loss
Keywords: Cochlear implant; telerehabilitation; telecoaching
MeSH Terms: conditions — Hearing Loss | interventions — Telerehabilitation

STUDY DESIGN:
Intervention Model Description: Two groups of cochlear implanted children one group will take sessions online (case group) and the other group will take sessions face to face (control group)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation group (Active Comparator): Group of cochlear implanted children who will take sessions online by the Arabic online program that will be designed
  Interventions: Behavioral: Telerehabilitation and telecoaching
- Face to Face group (Placebo Comparator): Group of cochlear implanted children who will take sessions face to face in the classical way (control group)
  Interventions: Behavioral: Face to Face Language sessions

INTERVENTIONS:
Behavioral: Telerehabilitation and telecoaching — Language Sessions online and coaching parents online to improve language and social outcomes of their children
  Other Names: Teletherapy
  Arms: Telerehabilitation group
Behavioral: Face to Face Language sessions — Language sessions Face to Face at sohag phoniatrics unit
  Arms: Face to Face group

SUMMARY:
Design online program for language sessions for cochlear implanted children in arabic and monitor its validity and reliability to improve language outcome

DETAILED DESCRIPTION:
Design online program for teletherapy and coach parents to improve language of their children with cochlear implant and evaluate language outcome before and after teletherapy and compare it with control group who will take classical face to face sessions

ELIGIBILITY:
Inclusion Criteria:

* Cochlear implanted children with non verbal intelligence quotient 80 or above
* parents are compliant to the sessions

Exclusion Criteria:

* cochlear implanted children who have non verbal intelligence quotient less than 80 using the Arabic version of Stanford Binet intelligence scale 5th edition
* parents are non compliant to sessions

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2022-02 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
changes at Sohag university hospital protocol for hearing impaired children | changes from Before sessions and after 3months and 6months of sessions
  Measurement of changes at receptive (0 - 94) and expressive (0-94) language scores and auditory score (0 - 28) higher scores means better outcomes (El-Adawy et al., 2020)
changes at Preschool language scale four | changes from Before sessions and after 3 months and 6 months of sessions
  changes at Receptive raw score (0-62) and expressive language raw score (0-71) and total raw score (0-133) and receptive standard score (43-106), expressive standard score (42-115) and total standard score (55- 115) higher scores means better outcomes (El Sady et al., 2011)

SECONDARY OUTCOMES:
changes at the Arabic version of Stanford Binet intelligence scale fifth edition (Faraj, 2010) | changes from Before sessions and after 6 months of sessions
  Intelligence quotient measure score (50- 160) higher scores means better outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Ahlam AN Eladawy, professor, Study Chair — Sohag University; Ahmed EA Gelany, lecturer, Study Director — Sohag University; Hadeel E Awad, ass.lecturer, Principal Investigator — Sohag University
Locations (1):
- Sohag University, Sohag, Faculty of Medicine, Egypt

IPD SHARING:
Plan to Share IPD: Yes
study protocol
Supporting Information: Study Protocol
Time Frame: january 2026 to june 2026
Access Criteria: emailing the principal investigator

REFERENCES:
- [Background] El-Adawy, A., Emam, A., Mostafa, E., Gelaney, A. & Awad, H. (2020): Assessment protocol for Auditory and Language Abilities in Cochlear Implanted Children used in Sohag university hospital. Egyptian Journal of Neck Surgery and Otorhinolaryngology, 6(1), 17-36.
- [Background] El-Sady, S.R., El-Shoubary, A.M., Hafez, G.N. & Abo-Hasseba, A.M. (2011): Translated, modified and standardized Preschool Language Scale [Unpublished Thesis]. 4th ed. Cairo: Ain Shams Medical School.
- [Background] Faraj, S., (2010): Stanford-Binet Intelligence Scales (SB5), Fifth Edition. Cairo: the Anglo Egyptian Bookshop.